CLINICAL TRIAL: NCT05138640
Title: Prospective Evaluation of Bone Strength, Physical Activity, Falls, Subsequent Fractures and Mortality in Patients Presenting With a Recent Clinical Fracture
Brief Title: Bone Strength and Physical Activity in Patients With a Recent Clinical Fracture
Status: Completed | Type: Observational
Sponsor: Joop P.W. van den Bergh (Other)
Responsible Party: Sponsor-Investigator, Joop P.W. van den Bergh, Clinical Professor, VieCuri Medical Centre
Organization: VieCuri Medical Centre (Other)
Other Study IDs: NL45707.072.13
Record Dates: First submitted 2014-09-26; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Fractures, Bone; Patient Fall; Osteoporosis; Physical Activity
MeSH Terms: conditions — Fractures, Bone; Osteoporosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Not applicable. The study is designed as an observational cohort study — Not applicable. The study is desigend as an observational cohort study

SUMMARY:
The risk for a subsequent fracture is significantly higher in patients presenting with a fracture compared to individuals without a previous fracture and is highest within the first 2 years after the initial fracture. The risk for a subsequent fracture is not dependent of BMD as measured by conventional DXA. In recent studies, it has been shown that HRpQCT measurements provide information about bone structure, bone quality and bone strength in addition to BMD measurements. Diagnostic strategies should be focussed on bone quality and bone strength and fall prediction in the patients at high risk for falls, subsequent fracture and mortality such as patients with a recent fracture. Therefore, the investigators conduct a prospective observational study in 500 patients aged 50 years and older who present with a clinical fracture for evaluation of bone strength, physical activity, falls, subsequent fractures and mortality during a follow-up period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years and older with a recent fracture that is being evaluated at the FLS at VieCuri MC.
* Patients who understand the conditions of the study and are willing and able to comply with the scheduled biochemical study procedures
* Patients who signed the Ethics Committee approved specific Informed Consent Form prior to inclusion.

Exclusion Criteria:

* Patients with malignancy metastatic to the bone.
* Patients with osteomyelitis.
* Patients with fractures due to failure of a prosthesis.
* Patients, who as judged by the Principal Investigator, are mentally incompetent. Patients who are compos mentis and understand the patient information, will not be considered mentally incompetent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a recent fracture evaluated at the FLS at VieCuri MC Venlo
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-10; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Bone strength assessed with HRpQCT | 3 years
  Difference in bone strength, estimated by micro-finite element analyses, will be compared between patients with and without a subsequent fracture within 3 years of follow-up.

SECONDARY OUTCOMES:
Subsequent falls within 3 years after a fracture | 3 years
  Number of patients sustaining a new fall during 3 years of follow-up.
Mortality | 3 years
  Number of patients deceased during 3 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: J PW van den Bergh, MD, PhD, Principal Investigator — VieCuri Medical Centre
Locations (1):
- VieCuri Medical Centre, Venlo, Limburg, Netherlands